CLINICAL TRIAL: NCT05143502
Title: Role of Montelukast in the Management of Chronic Rhinosinusitis With Nasal Polyps.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Aldein Samir Abd Elazeem Mohammed, Residant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Montelukast in nasal polyps
Record Dates: First submitted 2021-10-08; First posted 2021-12-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Montelukast; Chronic Rhinosinusitis With Nasal Polyps
Keywords: Montelukast; Chronic Rhinosinusitis with Nasal Polyps
MeSH Terms: interventions — montelukast; Prednisolone; fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Montelukast Group (Experimental): Patients in group A (interventional group) will be treated with fluticasone furoate nasal: (50 micrograms /spray ) 100 micrograms (2 sprays) in each nostril twice daily plus oral montelukast (montelukast 10 mg, once a day) for 3 monthes and oral Prednisolone 40 mg/day for two weeks.
  Interventions: Drug: Montelukast; Drug: Prednisolone; Drug: Fluticasone Furoate
- Control Group (Active Comparator): Subjects in treatment group B will receive topical and systemic steroids in an identical regimen only.
  Interventions: Drug: Prednisolone; Drug: Fluticasone Furoate

INTERVENTIONS:
Drug: Montelukast — Montelukast is a leukotrienes antagonist which has proven efficacious in chronic inflammatory conditions of the airways, including allergic rhinitis, asthma, and aspirin-exacerbated respiratory disease (AERD), all diseases that often coexist with CRSwNP.
  We will use oral Montelukast (montelukast 10 mg, once a day) for 3 monthes
  Arms: Montelukast Group
Drug: Prednisolone — Oral Prednisolone 40 mg/day for two weeks.
Drug: Fluticasone Furoate — fluticasone furoate nasal: (50 micrograms /spray ) 100 micrograms (2 sprays) in each nostril twice daily

SUMMARY:
The aim of the work is to examine the efficacy of montelukast as an adjunct to steroid therapy in patients with chronic rhinosinusitis with nasal polyps.

DETAILED DESCRIPTION:
Population and Methods The study will be conducted at the otorhinolaryngology department in Assiut University Hospital.

* Study design: prospective randomized controlled trial.
* .
* Methodology:

After fulfilling all inclusion and exclusion criteria all patients will be subjected to

A. Full history taking including :

1. Personal History
2. History of sinonasal symptoms (nasal obstruction, nasal discharge, headache, hyposmia, sneezing, itching, facial pain…etc)
3. History of nasal surgery.
4. Other ENT symptoms
5. General symptoms suggestive of atopy
6. History of general medical illness.

B. Examination :

* 1. General examination.
* 2. Full ENT examination.
* 3. Nasal endoscopy.

C. Investigations :

Multi-slice computer tomography (MSCT) of nose and paranasal sinuses axial, coronal and sagittal cuts without contrast .

D. Management :

Patients will be divided into 2 equal groups. Patients in group A will be treated with fluticasone furoate nasal: (50 micrograms /spray ) 100 micrograms (2 sprays) in each nostril twice daily plus oral montelukast (montelukast 10 mg, once a day) for 3 monthes and oral Prednisolone 40 mg/day for two weeks. Subjects in treatment group B will receive topical and systemic steroids in an identical regimen only.

.

ELIGIBILITY:
Inclusion Criteria:

* - 1- Adult patients (aged 18 years and over)
* 2- Bilateral denovo nasal polyps confirmed by nasal endoscopy and CT scan.

Exclusion Criteria:

* - 1- CRS patients without nasal polyposis.
* 2- Patient with unilateral nasal polyp.
* 3- Revision cases (history of previous surgical treatment).
* 4- Patient with fungal rhinosinusitis..
* 5- Pregnancy and lactation.
* 6- Malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change at nasal polyp size | after 12 weeks from the start of treatment
  Each CRSwNP patient will undergo nasal endoscopy to score the polyp size (0-4) in both nasal cavities using a modified Lildholdt scoring system:
  0 = no nasal polyps.
  1. small nasal polyps not reaching the inferior border of the middle turbinate.
  2. nasal polyps reaching beyond the inferior border of the middle turbinate.
  3. large nasal polyps reaching the lower edge of the inferior turbinate
  4. very large nasal polyps in contact with the floor of the nasal cavity.

SECONDARY OUTCOMES:
Nasal symptoms. | after 12 weeks from the start of treatment
  All participants will asked to score five sinonasal symptoms (nasal congestion/obstruction, anterior rhinorrhea, posterior rhinorrhea, loss of smell, and facial pain) from 0 to 4.
  0 = symptom-free/no symptom.
  1. mild symptom.
  2. moderate symptom.
  3. severe symptom.
  4. very severe symptom. This score will be assessed at the screening visit and follow-up visits at 4, 8 and 12 weeks. The total five-symptom score (T5SS) obtained with the sum of the individual symptoms (0-20).
Radiological evaluation | after 12 weeks from the start of treatment
  CT scan of the nose and paranasal sinuses will performed to all patients before and after the treatment and staged using the Lund-Mackay (LMK) scoring system where each sinus (maxillar, anterior ethmoidal, posterior eth-moidal, frontal, esphenoidal) is scored for opacification (0, no opacity; 1, partial opacity; 2, total opacity), and the ostiomeatal complex is scored 0 (no obstruction) or 2 (obstruction). The uni-lateral score goes from 0 to 12 whereas the bilateral score goes from 0 to 24.
Quality of life score | after 12 weeks from the start of treatment
  Subjects will complete validated questionnaire related to general quality of life lCSD (International Classification of Sinus Disease) before and after treatment. The ICSD records patients' symptoms of facial pain and pressure; headache ;nasal blockage Or congestion; nasal discharge; disturbance of smell; and Over all discomfort on a 0 to 10 ordinal scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Langdon C, Mullol J. Nasal polyps in patients with asthma: prevalence, impact, and management challenges. J Asthma Allergy. 2016 Mar 14;9:45-53. doi: 10.2147/JAA.S86251. eCollection 2016. PMID 27042129
- [Background] Johansson L, Akerlund A, Holmberg K, Melen I, Bende M. Prevalence of nasal polyps in adults: the Skovde population-based study. Ann Otol Rhinol Laryngol. 2003 Jul;112(7):625-9. doi: 10.1177/000348940311200709. PMID 12903683
- [Background] Wang X, Zhang N, Bo M, Holtappels G, Zheng M, Lou H, Wang H, Zhang L, Bachert C. Diversity of TH cytokine profiles in patients with chronic rhinosinusitis: A multicenter study in Europe, Asia, and Oceania. J Allergy Clin Immunol. 2016 Nov;138(5):1344-1353. doi: 10.1016/j.jaci.2016.05.041. Epub 2016 Jul 15. PMID 27544740
- [Background] Scadding GK, Durham SR, Mirakian R, Jones NS, Drake-Lee AB, Ryan D, Dixon TA, Huber PA, Nasser SM; British Society for Allergy and Clinical Immunology. BSACI guidelines for the management of rhinosinusitis and nasal polyposis. Clin Exp Allergy. 2008 Feb;38(2):260-75. doi: 10.1111/j.1365-2222.2007.02889.x. Epub 2007 Dec 20. PMID 18167126
- [Background] Joe SA, Thambi R, Huang J. A systematic review of the use of intranasal steroids in the treatment of chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2008 Sep;139(3):340-7. doi: 10.1016/j.otohns.2008.05.628. PMID 18722209
- [Background] Rudmik L, Schlosser RJ, Smith TL, Soler ZM. Impact of topical nasal steroid therapy on symptoms of nasal polyposis: a meta-analysis. Laryngoscope. 2012 Jul;122(7):1431-7. doi: 10.1002/lary.23259. Epub 2012 Mar 12. PMID 22410935
- [Background] Fokkens W, Desrosiers M, Harvey R, Hopkins C, Mullol J, Philpott C, Alobid I, Anselmo-Lima WT, Bachert C, Baroody F, Bernal-Sprekelsen M, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Douglas R, Gevaert P, Hafner A, Hellings P, Joos G, Kalogjera L, Kern R, Knill A, Kocks J, Landis BN, Limpens J, Lebeer S, Lourenco O, Matricardi PM, Meco C, O Mahony L, Reitsma S, Ryan D, Schlosser R, Senior B, Smith T, Teeling T, Tomazic PV, Toppila-Salmi S, Wang DY, Wang D, Zhang L, Lund V. EPOS2020: development strategy and goals for the latest European Position Paper on Rhinosinusitis. Rhinology. 2019 Jun 1;57(3):162-168. doi: 10.4193/Rhin19.080. PMID 30810118
- [Background] Holgate ST, Peters-Golden M, Panettieri RA, Henderson WR Jr. Roles of cysteinyl leukotrienes in airway inflammation, smooth muscle function, and remodeling. J Allergy Clin Immunol. 2003 Jan;111(1 Suppl):S18-34; discussion S34-6. doi: 10.1067/mai.2003.25. PMID 12532084
- [Background] Cao Y, Wang J, Bunjhoo H, Xie M, Xu Y, Fang H. Comparison of leukotriene receptor antagonists in addition to inhaled corticosteroid and inhaled corticosteroid alone in the treatment of adolescents and adults with bronchial asthma: a meta-analysis. Asian Pac J Allergy Immunol. 2012 Jun;30(2):130-8. PMID 22830292